CLINICAL TRIAL: NCT03154814
Title: High-dose Ulinastatin Improves Postoperative Oxygenation in Patients Undergoing Aortic Valve Surgery With Cardiopulmonary Bypass
Brief Title: Ulinastatin Improves Postoperative Oxygenation After Cardiopulmonary Bypass
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH1160051
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cardiopulmonary Bypass; Cardiac Surgery
Keywords: ulinastatin; cardiopulmonary bypass; cardiac surgery
MeSH Terms: interventions — urinastatin

STUDY DESIGN:
Intervention Model Description: Retrospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ulinastatin treatment (Experimental): ulinastatin (10000 U/kg and 5000 U/kg/h) was administered during CPB
  Interventions: Drug: ulinastatin
- control (Placebo Comparator): conventional CPB was applied without ulinastatin treatment
  Interventions: Drug: control

INTERVENTIONS:
Drug: ulinastatin — ulinastatin (10000 U/kg and 5000 U/kg/h) was administered during CPB
  Other Names: ulinastatin administration
  Arms: ulinastatin treatment
Drug: control — conventional CPB was applied without ulinastatin treatment
  Other Names: placebo
  Arms: control

SUMMARY:
Retrospective study determine whether ulinastatin enhances postoperative pulmonary oxygenation after cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
This retrospective study evaluate patients who underwent aortic valvular surgery under moderate hypothermic CPB. The patients were classified into two groups: patients in whom high-dose ulinastatin (10,000 U/kg and 5,000 U/kg/h) was administered during CPB (Group-U); and patients in whom ulinastatin was not administered (Group-C). We measured PaO2/FiO2 at the following time points: before CPB (Pre-CPB), 2 hours after weaning from CPB (Post-CPB) and within 6 hours after admission to the ICU. The lengths of ventilator care and ICU stay were also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent aortic repair or replacement under moderate hypothermic CPB

Exclusion Criteria:

* Preoperative:

< 19 years old, > 85 years old, emergency operation, reoperation, left ventricular ejection fraction < 50%, arrhythmia, ischaemic myocardial disease, uncontrollable hypertension or hypotension, pericardial disease, pre-existing hepatic dysfunction, pre-existing renal dysfunction or underlying lung disease.

* Intraoperative:

intraoperative application of an intra-aortic balloon pump, administration of steroids or tranexamic acid, and transfusion of fresh frozen plasma or platelet concentrates during CPB.

* Postoperative:

reoperation for surgical correction of intractable postoperative bleeding within 2 hours after the end of surgery and transfusion of any banked blood products.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
change of arterial oxygen partial pressure (PaO2)/fraction of inspired oxygen (FiO2) during CPB | before CPB (Day 0), 2hours after CPB(Day 0), within 6hour after admission to intensive care unit(Day 0)
  pulmonary oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Tae-yop Kim, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes